CLINICAL TRIAL: NCT04231396
Title: Effects of Audiobooks for Hearing Loss App as Auditory Training for Those With CI and HA Users.
Brief Title: Audiobooks for Hearing Loss App as Auditory Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioSpeech (Industry)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Kirsty Lindaas-Hamilton, Principal Investigator, BioSpeech
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R44DC017403-01A1 (NIH)
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Results first posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Hearing Loss; Hearing Impaired Children; Hearing Impairment
MeSH Terms: conditions — Hearing Loss | interventions — Sound Recordings

STUDY DESIGN:
Intervention Model Description: 40 subjects will participate in total, including children and adults with HL aided with either Hearing Aids or Cochlear Implants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HA and CI Users using Audiobooks for Hearing Loss for Auditory Training (Other): study participants will be seen weekly for 12 weeks and will use the Audiobooks for HL App for the final 6 weeks using the App at least two hours per week on their own. The researcher will conduct 12 weekly in-home visits where the following will be done:
  First 6 weeks:
  • Partial BKB-SIN will be administered
  Final 6 weeks:
  * Partial BKB-SIN will be administered
  * Conduct a comprehension test.
  * Address any usability issues the participant brings up.
  * Review and set new weekly goals Final session: Conduct Final Usability survey
  Interventions: Other: Audiobooks for hearing loss App

INTERVENTIONS:
Other: Audiobooks for hearing loss App — Same as Arm 1

SUMMARY:
The goal of the proposed project is to create an Audiobooks for Hearing Loss (HL) App - an audiobook App that has a wide array of user-selectable features designed to provide auditory training. The effects of the Audiobooks for Hearing Loss App as Auditory Training for those With CI and HA Users was measured with a 6-week trial of using the app and measuring changes in listener abilities and adherence to the program.

DETAILED DESCRIPTION:
Twenty percent or more Americans have a Hearing Loss (HL), a commonly used term that includes congenital deafness as well as aging-related hearing challenges, so severe that it may make communication difficult. Worldwide, this translates into 65 million people with English as a first language.

Hearing aids (HAs) and cochlear implants (CI's) are not enough to remedy this. The types of enhancement these devices can perform is inherently limited due to the requirement that they need to perform their task in real time, since otherwise they would not be lip-synchronized, which is essential in face-to-face communication. For example, they cannot change the temporal structure of incoming speech, even if that may help intelligibility. But there is a deeper shortcoming. When individuals wait too long with obtaining these devices, synaptic and pathway re-organization takes place in the auditory cortex that needs to be addressed, and mere device usage may not be up to this task. Cochlear implants provide a special challenge: Individuals may initially have great difficulty deciphering the unfamiliar sensory input generated by these devices.

There is a growing consensus that HL cannot be addressed with HAs or CIs alone: auditory training is also needed. While face-to-face auditory training is available, this intervention is generally not covered by insurance plans. Auditory training Apps have become available to fill this need in a cost-effective manner. Unfortunately, evidence for the efficacy of these products is weak; a recent large-scale randomized controlled trial found no effect on a wide range of outcome measures. A likely suspect for these results is that most aural rehab Apps are repetitive, even with gamification and rewards. A popular method used by individuals with HL to improve their listening skills is listening to audiobooks. Audiobooks have the strong advantage over many aural rehab Apps of being intrinsically motivating. However, existing audiobooks do not adequately accommodate individuals with more severe levels of HL unless they are fundamentally re-thought.

The goal of the proposed project is to create an Audiobooks for Hearing Loss (HL) App - an audiobook App that has a wide array of user-selectable features designed to provide auditory training: Help individuals with recent Cochlear Implants/Hearing Aids through the difficult initial adjustment process, and help with transitioning at one's own pace toward the goal of understanding "habitual speech" (speech spoken without special effort to be intelligible). Even if not used for auditory training, this app would provide access to audiobooks where standard audiobooks fail. Thus, the App serves both auditory training and accessibility. Proposed features include enhanced ("clear") speech modes, visual support by simultaneous display of text and a talking face, and other features that can be enabled or disabled to serve the user's unique needs.

ELIGIBILITY:
Inclusion Criteria:

*Because of the COVID-19 Pandemic and low enrollment numbers for certain HL subgroups in the study, the effectiveness of the Audiobooks for Hearing Loss App was measured for the overall group.

Participants had to fall into one of the following five HL subgroups: (1) Adults with HA, moderate HL (41-55 dB); (2) Adults with HA, moderately-severe to severe HL (56 to 90 dB); (3) Adults with non-recent CI, post-lingually deaf; (4) Children, ages 9+, non-recent CI, pre-lingually deaf; and (5) Adults and Children, ages 9+, recent CI, post-lingually deaf. These five subgroups span broad ranges in terms of: (1) age (adults vs. children); (2) severity of hearing loss; (3) device used (HAs vs. Cis); (4) familiarity with device (recent vs. longer-term); and (5) onset of HL (pre-lingual vs. post-lingual. The team expects the highest efficacy for children and adults with recent CI who are post-lingually deaf; the lowest efficacy for adults with HA with either moderate of severe HL; and intermediate efficacy for children with non-recent CI who are pre-lingually deaf.

* speaking English as first language,
* and being able to read at least a first-grade level.

Exclusion Criteria:

* no suspicions of cognitive deficits or vision impairments that would interfere with system usage or invalidate usability assessment,
* no signs of external ear disease,
* and all participants will be tested with the Expressive One-Word Picture Vocabulary Test, 4th Edition (EOWPVT-4; Brownell 2000), normed for ages of 2 and older, and are required to score in the 15th percentile or better.

Ages: 9 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2021-09-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- OHSU, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The COVID-19 pandemic impacted recruitment efforts. Participants were recruited by flyers and posted at multiple sources, including local healthcare specialists (Audiologist and Otolaryngologist offices), schools, and hearing loss support group meetings. Participants were recruited via Facebook ad on Hospitals' Facebook Pages. Recruitment occurred between February 2021 and June 2021. The first participant enrolled on February 25, 2021 and the last participant enrolled on June 23, 2021.
Groups:
- HA and CI Users Using Audiobooks for Hearing Loss App as Auditory Training: *The COVID-19 Pandemic and low enrollment numbers for certain HL subgroups in the study caused an imbalance of subgroup numbers for comparisons, therefore, the effectiveness of the Audiobooks for Hearing Loss App was measured for the overall group.
  Study participants were seen for 12 weeks and used the Audiobooks for HL App for the final 6 weeks using the App at least two hours per week on their own. The researcher conducted 12 weekly visits where the following was done:
  First 6 weeks:
  • Administer partial BKB-SIN test
  Final 6 weeks:
  * Administer partial BKB-SIN test
  * Conduct a comprehension test.
  * Address any usability issues the participant brings up.
  * Review and set new weekly goals Final session: Conduct Final Usability survey
Period: Overall Study
Arm/Group | HA and CI Users Using Audiobooks for Hearing Loss App as Auditory Training
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- HA and CI Users Using the Audiobooks for Hearing Loss App as Auditory Training: *The COVID-19 Pandemic and low enrollment numbers for certain HL subgroups in the study caused an imbalance of subgroup numbers for comparisons, therefore, the effectiveness of the Audiobooks for Hearing Loss App was measured for the overall group.
  Study participants were seen for 12 weeks and used the Audiobooks for HL App for the final 6 weeks using the App at least two hours per week on their own. The researcher conducted 12 weekly visits where the following was done:
  First 6 weeks:
  • Administer partial BKB-SIN test
  Final 6 weeks:
  * Administer partial BKB-SIN test
  * Conduct a comprehension test.
  * Address any usability issues the participant brings up.
  * Review and set new weekly goals Final session: Conduct Final Usability survey
Arm/Group | HA and CI Users Using the Audiobooks for Hearing Loss App as Auditory Training
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 10
  >=65 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 27
Region of Enrollment [Number; unit: participants]
  United States | 27
Hearing Loss resulting in: HA or CI [Count of Participants; unit: Participants] | 27

OUTCOME MEASURES:

1. Primary Outcome: Audiobooks Efficacy: Change in Slope of Curve for SNR Loss Scores on a Scale/Week for Partial BKB-SIN Hearing Test
Description: Speech in noise test; partial BKB-SIN hearing test. SNR Loss scores based on normative sample data on decibel (dB) measures. where Minimum value is 0 dB, Maximum value 15+ dB. Lower scores mean better outcome, 0-3dB = hearing normal; 3-7 dB = Mild SNR loss; 7-15 dB = Moderate SNR loss; >15 db = Severe SNR loss. Slopes of BKB-SIN (Background Noise partial tests) were measured from the Auditory Training portion of the study: weeks 7-12. We used a smoothing method for statistical analysis: isotonic regression (isoreg(), via R). This method is the fundamental assumption that the scores of these 6 weeks will be non-increasing indicating better outcome; improved listening scores on the BKB-SIN partial tests.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale/week
Groups:
- HA and CI Users Using the Audiobooks for Hearing Loss App as Auditory Training: Study participants will use the Audiobooks for HL App for 12 weeks using the App at least two hours per week on their own. The researcher will conduct 12 weekly visits where the following will be done:
  First 6 weeks:
  • Partial BKB-SIN will be administered
  Final 6 weeks:
  * Partial BKB-SIN will be administered
  * Conduct a comprehension test.
  * Address any usability issues the participant brings up.
  * Review and set new weekly goals Final session: Conduct Final Usability survey of the App
Arm/Group | HA and CI Users Using the Audiobooks for Hearing Loss App as Auditory Training
Number analyzed (Participants) | 27
units on a scale/week
  week 7 | 5.978 (.712)
  week 8 | 5.889 (.716)
  week 9 | 5.757 (.720)
  week 10 | 5.600 (.711)
  week 11 | 5.398 (.708)
  week 12 | 5.088 (.725)
Statistical Analysis 1: Comparison: HA and CI Users Using the Audiobooks for Hearing Loss App as Auditory Training; The SNR Loss scores computed the means per client and week (1-12), with a smoothing method: isotonic regression (isoreg, via R). The slopes (lsfit, via R) calculated of the smoothed means separately per client, per 7-9 weeks (early training weeks), and per 10-12 weeks (final training weeks). This created slope differences, per client; Test type: Superiority; p = .037, t-test, 1 sided; Mean Difference (Final Values) = .1456, 95% CI 2-sided [.012 to .279]

2. Secondary Outcome: Audiobooks Positive Responses: Percentage of Positive Responses to Final Usability Survey Question: Would You Buy or Recommend Audiobooks for HL App as Auditory Training
Description: Percentage of positive answers on Final Usability Survey: "Would you buy or recommend the Audiobooks for Hearing Loss App for yourself or someone you know who recently got a new Hearing Aid or Cochlear Implant." Clients filled out final usability survey at end of 12-week study.
Time Frame: 6 weeks
Measure: Number; unit: percentage of positive answers
Groups:
- HA and CI Users Using the Audiobooks for Hearing Loss App as Auditory Training: study participants will use the Audiobooks for HL App for 12 weeks using the App at least two hours per week on their own. The researcher will conduct 12 weekly visits where the following will be done:
  First 6 weeks:
  • Partial BKB-SIN will be administered
  Final 6 weeks:
  * Partial BKB-SIN will be administered
  * Conduct a comprehension test.
  * Address any usability issues the participant brings up.
  * Review and set new weekly goals Final session: Conduct Final Usability survey
Arm/Group | HA and CI Users Using the Audiobooks for Hearing Loss App as Auditory Training
Number analyzed (Participants) | 27
percentage of positive answers | 77

3. Secondary Outcome: Audiobooks Adherence: Overall Mean Score of Weekly Goals Met for HA and CI Users Using the Audiobooks for HL App as an Auditory Training Program
Description: Meeting specific weekly goals (yes/no) for using the Audiobooks for HL App with was a measure of adherence to this Auditory Training program. Researcher tracked whether HA and CI Users met their weekly goals during weekly check-ins. The researcher recorded information from the App's dashboard about whether the client had met the previous week's goals. The dashboard shows the Client's weekly goals of: Minutes of listening, minutes of listening in Standard Speech, minutes of Pure Listening (audio only), minutes of no text support, minutes of listening in background noise. New goals were updated for the upcoming week with increased difficulty based on goal performance.
  The scale used for the overall mean scores reported is 0 to 1.0 where the minimum value is 0 and maximum value is 1. Computing in percentage 0 = 0% for meeting that specific goal and 1.0 = 100% for meeting that specific goal, so higher scores closer to 1.0 mean greater adherence to this Auditory Training program.
Time Frame: 6 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | HA and CI Users Using the Audiobooks for Hearing Loss App as Auditory Training
Number analyzed (Participants) | 27
score on a scale
  Minutes of listening, met goal of 2 hours | .9275 (.1313)
  Minutes of Standard Speech, met goal | .9667 (.0680)
  Minutes of Pure Listening, met goal | .9545 (.0917)
  Minutes of not text support, met goal | .9420 (.1190)
  Minutes of listening in background noise, met goal | .9815 (.0539)

ADVERSE EVENTS:
Time Frame: 6 months; during the overall period of the study while clients were seen: February 2021-September 2021
Description: The anticipated potential adversity inherent in this study is minimal. Process for identifying AEs and SAEs will be to have the researcher document information regarding if any events occur at each weekly visit using the adverse event form. Then the researcher will promptly report the AEs and/or SAEs to the study PI (and beyond, as required). Alexandra Dimitrova, MD, MA, MCR, an Assistant Professor of Neurology at OHSU will serve as the Independent Safety Monitor (ISM).
Arm/Group | HA and CI Users Using the Audiobooks for Hearing Loss App as Auditory Training
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

LIMITATIONS AND CAVEATS:
COVID-19 impacted enrollment causing an imbalance of subgroup numbers for comparisons, so the effectiveness of the Audiobooks was measured for the overall group.

The partial BKB-SIN hearing test that was given weekly consisted of 4 lists of sentences vs. the comprehensive BKB-SIN hearing test, which is comprised of 36 lists of sentences. The smaller sample size; number of items used on the partial BKB-SIN hearing test often produced significant variability which can lead to unreliable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/96/NCT04231396/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/96/NCT04231396/ICF_001.pdf